CLINICAL TRIAL: NCT05682963
Title: Effect of Square- Stepping Exercises on Mobility, Balance and Knee Joint Position Sense in Individuals With Multiple Sclerosis
Brief Title: Efficacy of Square- Stepping Exercises in Individuals With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, müge içelli, lecturer, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PU-FTR-MI-01
Record Dates: First submitted 2022-12-24; First posted 2023-01-12 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Mobility; Balance; Position Sense
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Total of two groups: Square stepping exercise program group and home exercise program group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Square-Stepping Exercise Program Group (Active Comparator): Square stepping exercise is performed on a thin exercise mat divided into 40 small squares of 250 cm x 100 cm. Participants practice a set of step patterns on the mat. Square step exercises are a low-cost, highly accessible and fun exercise method. It is known that it improves motor performance and muscle strength in healthy young individuals, and has positive effects on functional fitness and gait parameters in individuals with osteoarthritis. It is known to have positive effects on balance, fall risk, walking ability, physical and cognitive function in elderly individuals. It will be applied to examine the effects on mobility, balance and position sense in individuals with multiple sclerosis.
  Interventions: Other: Square Step Exercises Program
- Home Exercise Program Group (Active Comparator): The home exercise program group will implement a protocol of frenkel's coordination exercises developed for balance and coordination therapy. The exercise protocol, which includes frenkel's coordination exercises, will be delivered to the patient in the form of a brochure and in the form of a Compact Disc (CD) with video images.
  Interventions: Other: Home Exercise Program

INTERVENTIONS:
Other: Square Step Exercises Program — Intervention description: patient will be treated for eight weeks, two days a week, one session a day, and total 16 session. Each session will be 45 minute.
  Arms: Square-Stepping Exercise Program Group
Other: Home Exercise Program — Frenkel's coordination exercises will be applied as a home program for 8 weeks, 2 days a week, with each exercise session 15-30 minutes excluding rest periods.
  Arms: Home Exercise Program Group

SUMMARY:
Square stepping exercises can promote correct foot placement, fast and coordinated step patterns, and sensory-motor interaction. The aim of this study is to examine the effect of square stepping exercises on mobility, balance and knee joint position sense in individuals with multiple sclerosis.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic, inflammatory, autoimmune disease of the central nervous system that results in neurological disability. Complex gene-environment interactions play a role in the etiology of multiple sclerosis. Multiple sclerosis is more common in women than men, with a ratio ranging from 2:1 to 3:1.

MS is a very heterogeneous disease and it can have very variable clinical signs and symptoms, including motor, sensory, autonomic and cognitive disorders, depending on the region of the central nervous system. Balance and mobility disorders are the leading symptoms of MS. In addition, somatosensory disorders are frequently encountered as the initial symptom. Disorders in position sense, which is one of the components of somatosensory sense, is an important determinant of limitations during dynamic activities such as walking and balance. In order to reduce disability and improve function in individuals with Multiple Sclerosis, square stepping exercises protocol will be given to one group and a home exercise program protocol to the other group. Created by Shigematsu and Okura to improve balance and reduce the risk of falling, the square stepping exercises is performed on a thin exercise mat divided into 40 small squares of 250 cm x 100 cm. There are a number of step patterns that must be followed by the participants. Certain step patterns will be repeated 3-5 times to the participants and the participant will be asked to repeat the same pattern. As a home exercise protocol, a program consisting of frenkel exercises developed by Professor Heinrich Sebastian Frenkel for the treatment of gait, balance and coordination will be applied.

Square stepping exercises can promote correct foot placement, fast and coordinated step patterns, and sensory-motor interaction. The aim of this study is to examine the effect of square stepping exercises on mobility, balance and knee joint position sense in individuals with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Having a disability score of less than 4
* Being between 20-50 years old
* Not having an attack in the last month
* Patients without lower extremity spasticity according to Modified Ashworth Scale (MAS)

Exclusion Criteria:

* Having a neurological disease other than Multiple Sclerosis
* Having an Multiple Sclerosis attack during the study
* Having had orthopedic surgery affecting balance
* Presence of cognitive and psychiatric influences that will affect participation in the study
* Having a cardiovascular or pulmonary history that would inhibit participation in the study
* Have received steroid and/or immunosuppressive therapy in the past four weeks

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Timed 25-Foot Walk (T25-FW) Test | 8 weeks
  With the Timed 25-Foot Walk (T25-FW) Test, the patient's walking speed and lower extremity functions are evaluated. The patient is asked to walk a distance of 7.62 m (25 feet) safely and as quickly as possible. The passing time is recorded in seconds with the chronometer. The T25-FW is the best-defined measurement method for the measurement of gait disturbance in patients with MS and the evaluation of gait speeds of patients with many gait disorders in the clinical setting.

SECONDARY OUTCOMES:
Five Times Sit to Stand Test | 8 week
  The patient is asked to sit down and stand up from a standard chair as fast as possible with 5 repetitions. The test starts from a sitting position and ends in a sitting position. The result is recorded in seconds. This method, which is valid and reliable in MS, has been shown to be associated with lower extremity muscle strength and balance. Low times are indicative of high performance.
Four Step Square Test (FSST) | 8 week
  It is a test method used to evaluate the dynamic balance status of individuals. Four squares are formed by placing two canes on a flat surface. All squares are numbered. At the beginning of the test, the patient is told to step into each square as fast as possible, without touching the canes, in consecutive order (2-3-4-1-4-3-2-1). (Requires the patient to step forward, backward, to the right and left side). The time to complete the test is recorded as a score. Low times are indicative of high performance.
Activity-Specific Balance Confidence Scale | 8 week
  It measures the effect of balance disorder on the psychology of the patient. It is a self-report scale in which patients evaluate how confidently they can perform 16 activities that require balance skills, both inside and outside the home, between 0% (unsafe) and 100% (with complete confidence).
Knee Joint Position Sense | 8 week
  The knee joint position sense will be evaluated with the KFORCE Sens® electrogoniometer. For standardization of sensory measurements, the patient is evaluated in a sitting position with the back supported and the hips and knees flexed to 90°. The knee extension angles of 30 and 60 degrees according to the initial position are determined as the target angle, and the repositioning error of the participant is checked. When the participant brings the knee joint to the target angle, the participant is asked to learn the angle by waiting five seconds at this point. Then the knee is brought to the neutral position and the patient is asked to find the target angle. For the target angles, the measurements are repeated three times, the average value is calculated and the reposition error degree of the patients is recorded.
Expanded Disability Status Scale (EDSS) | 8 week
  The EDSS scale is a scale that provides information about the disability status of the patient. Functional systems evaluated by EDSS are pyramidal, cerebral, cerebellar, visual, sensory, brain stem, bladder and bowel functions. Scoring is done between 0 and 10. Scoring between 0 and 3.5 indicates mild disability, scoring between 4.0 and 6.5 indicates moderate disability, and scoring between 7.0 and 10.0 indicates severe disability.

CONTACTS AND LOCATIONS:
Overall Officials: Müge İçelli, M.Sc., Principal Investigator — Pamukkale University Denizli Health Services Vocational School of Higher Education
Locations (1):
- Pamukkale University Denizli Health Services Vocational School of Higher Education, Denizli, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No